CLINICAL TRIAL: NCT00606658
Title: Usefulness of Shirodhara (Oil Dripping Treatment in Ayurveda) for Insomnia - A Case Series
Brief Title: Usefulness of Shirodhara for Insomnia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Southern California University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sivarama Vinjamury, Associate Professor, Southern California University of Health Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCU-07-VINJ002
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Insomnia
Keywords: Insomnia; Ayurveda; Shirodhara; Quality of Life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oil dripping therapy (Other): Single Arm
  Interventions: Procedure: Shirodhara Oil Treatment

INTERVENTIONS:
Procedure: Shirodhara Oil Treatment — Oil dripping on the forehead in a constant stream for about 40 minutes for five consecutive days.

SUMMARY:
This pilot study will attempt to test the effects of this non-invasive procedure on a small sample of insomnia patients and also determine the feasibility of recruiting and retaining participants during the trial for such treatments in the United States.

DETAILED DESCRIPTION:
A prospective case series design will be adopted. Due to the small sample size and the preliminary nature of the study, a single case study or case series are classified under Observational Descriptive Studies. The investigators will seek local Institutional Review Board (IRB) approval. Ten volunteers who respond to the recruitment efforts will be enrolled into the study. Successful enrollment is based on strict inclusion and exclusion criteria. Brahmi oil (sesame oil processed with Bacopa monieri and other herbs) will be used to perform Shirodhara. Each participant will be treated for 40 minutes for five consecutive days. Outcome measures data will be collected at baseline, third day and fifth day and a week after the treatment is over. Additionally, demographic data will be collected at baseline as well. Participants will be asked to record any adverse events or side effects they observe during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 of either sex
* Duration of insomnia at least one year
* Willing to sign an informed consent
* A score of minimum 14 on the Insomnia severity index

Exclusion Criteria:

* Comorbidities such as Depression or any other psychological conditions that require medications
* Currently on prescription medication for insomnia
* Serious medical conditions such as uncontrolled hypertension, uncontrolled diabetes, or any other acute condition that disturbs sleep and requires waking up in the middle of the night
* Participants unwilling to comply with the protocol
* Anyone who is in litigation or receiving disability, workers' compensation benefits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline, end of five days and end of 14 days

SECONDARY OUTCOMES:
HD-16 Quality of Life Scale | Baseline, end of 5 days and 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sivarama P Vinjamury, MAOM, Principal Investigator — Southern California University of Health Sciences
Locations (1):
- Southern California University of Health Sciences, Whittier, California, United States

REFERENCES:
- See also: Visit Southern California University of Health Sciences Website — http://www.scuhs.edu